CLINICAL TRIAL: NCT01071850
Title: A Phase 2, Double-Blind, Randomized, Placebo and Active-Controlled Dose-Finding Study to Assess the Efficacy, Safety and Tolerability of Multiple Oral Doses of ASP1941 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Effect of ASP1941 in Adult Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0004
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: ASP1941; Metformin; Type 2 diabetes; diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- ASP1941 lowest dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin
- ASP1941 low dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin
- ASP1941 high dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin
- ASP1941 highest dose (Experimental): oral tablet
  Interventions: Drug: ipragliflozin
- Metformin (Active Comparator): oral tablet
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): oral tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ipragliflozin — oral tablet
  Other Names: ASP1941
  Arms: ASP1941 high dose; ASP1941 highest dose; ASP1941 low dose; ASP1941 lowest dose
Drug: Metformin — oral tablet
  Arms: Metformin
Drug: Placebo — oral tablet
  Arms: Placebo

SUMMARY:
Evaluate the efficacy, safety, and tolerability of multiple doses of ASP1941 compared to placebo over 12 weeks of therapy in adult patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with type 2 diabetes
* Subject has a HbA1c value between 6.8 and 9.5%
* Subject has never, is not currently taking anti-diabetic medication OR is receiving a single anti- diabetic agent or low-doses two anti-diabetic medications and is willing to discontinue them during the study
* Subject is on a stable diet and exercise program
* Female subject is not pregnant and agrees to use an acceptable form of contraception throughout the duration of the study

Exclusion Criteria:

* Subject has type 1 diabetes mellitus
* Subject is using insulin therapy
* Subject has a serum creatinine higher than upper limit of normal
* Subject has an ALT and/or AST value higher than 3 times upper limit of normal or a total bilirubin value more than 2 times upper limit of normal
* Subject has persistent, uncontrolled severe hypertension as indicated by a

systolic blood pressure >180 mmHg or a diastolic blood pressure of

>110mmHg

* Subject has had significant cardiovascular disease such as myocardial infarction or a vascular intervention (e.g., angioplasty or stent) in the last 3 months
* Subject is known to have hepatitis or be a carrier of hepatitis B surface

antigen, hepatitis C virus antibody or is known positive for HIV1 and/or

HIV2

* Subject has a history of lactic acidosis
* Subject has a history of drug and alcohol abuse/dependency within last 12

months

* Subject has had a malignancy in the last 5 years, except for successfully

treated basal or squamous cell carcinoma of the skin or of the cervix

* Subject has a symptomatic urinary tract infection or genital infection
* Female subject is lactating
* Subject has an unstable medical or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2010-03-03 (Actual); Primary Completion 2011-04-11 (Actual); Study Completion 2011-04-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in Hemoglobin A1c (HbA1c) | 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline in fasting plasma glucose (FPG) | 12 weeks
Proportion of subjects achieving target goal of HbA1c <7.0% | 12 weeks
Proportion of subjects achieving target goal of HbA1c <6.5% | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (59):
- United States (37):
  - Parkway Medical Center, Birmingham, Alabama
  - Winston Technology Research, LLC, Haleyville, Alabama
  - Desert Clinical Research, Mesa, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Paul W. Davis, MD, PA, Pine Bluff, Arkansas
  - Clinical Innovations, Inc., Costa Mesa, California
  - Del Rosario Medical Clinic, Inc, Huntington Park, California
  - Torrance Clinical Research, Lomita, California
  - San Diego Managed Care Group Clinical Research, San Diego, California
  - Expresscare Clinical Research, Colorado Springs, Colorado
  - PAB Clinical Research, Brandon, Florida
  - Clinical Therapeutics Corp., Coral Gables, Florida
  - A.G.A Clinical Trials DBA Neostart Group, Hialeah, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - CSRA Partners in Health, Inc., Augusta, Georgia
  - Atlanta Vascular Research Foundation, Atlanta Cardiology & Primary Care P.C., Tucker, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - APEX Medical Research, AMR, Inc, Chicago, Illinois
  - MediSphere Medical Research, Evansville, Indiana
  - Bay West Endocrinology, Towson, Maryland
  - Prism Research, Saint Paul, Minnesota
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Rapid Medical Research, Cleveland, Ohio
  - Primecare of Southeastern Ohio, Inc., Zanesville, Ohio
  - Integris Family Care, Yukon, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Fleetwood Clinical Research, Fleetwood, Pennsylvania
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Southwind Medical Specialist, Memphis, Tennessee
  - Punzi Medical Center, Carrollton, Texas
  - Corpus Christi Family Wellness Center, Corpus Christi, Texas
  - Excel Clinical Research, LLC, Houston, Texas
  - Cetero Research, San Antonio, Texas
  - Aspen Clinical Research, Orem, Utah
- Colombia (6):
  - BIOMELAB, Barranquilla
  - Centro de Reumatologia y ortopedia, Barranquilla
  - Fundacion de Caribe para le Investigacion Biomedica, Barranquilla
  - Dexa Diad Servicios Medicos, Bogotá
  - School of Medicine University of Rosario, Bogotá
  - Fundacion Cardiovascular de Columbia, Floridablanca Santander
- India (6):
  - Diacon Hospital, Bangalore
  - Hormone Care and Research Centre, Ghaziabad
  - TOTALL Diabetes Hormone Institute Pvt.Ltd., Indore
  - S R Kalla Memorial Gastro & General Hospital, Jaipur
  - Bride, Bharti Hospital, Karnāl
  - Amrita Institute of Medical Sciences and Research Centre, AIMS, Kerala
- Mexico (6):
  - Unidad Metabólica y Cardiovascular, SC., Cuernavaca
  - Instituto Jaliscience de Investigacion Clinica, Guadalajara
  - Torre Medica Providencia, Guadalajara
  - Medical Care and Research, Mérida
  - CEDIME, Instituto Vascular, Mérida
  - Hospital Universitario Dr. Eleuterio Gonzalez, Monterrey
- Philippines (4):
  - Cebu Doctors' University Hospital, Cebu
  - St. Paul's Hospital, Iloilo City
  - Amang Rodriguez Memorial Medical Center, Marikina City
  - San Juan De Dios Hospital, Pasay

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- [Derived] Fonseca VA, Ferrannini E, Wilding JP, Wilpshaar W, Dhanjal P, Ball G, Klasen S. Active- and placebo-controlled dose-finding study to assess the efficacy, safety, and tolerability of multiple doses of ipragliflozin in patients with type 2 diabetes mellitus. J Diabetes Complications. 2013 May-Jun;27(3):268-73. doi: 10.1016/j.jdiacomp.2012.11.005. Epub 2012 Dec 29. PMID 23276620
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=1